CLINICAL TRIAL: NCT04561141
Title: Post Covid Syndrome: Clinical Pattern and Functional Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud, resident doctor, Assiut University
Other Study IDs: postcovid syndrome
Record Dates: First submitted 2020-09-22; First posted 2020-09-23 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim(s) of the Research :

1. Identify post covid symptoms
2. prevalance of post covid syndrome among survivours

DETAILED DESCRIPTION:
There is currently very limited information on the nature and prevalence of post-COVID-19 symptoms after hospital discharge. On 11th March 2020, corona virus disease 2019 (COVID-19) was declared a global pandemic by the World Health Organisation (WHO). Egypt has been one of the worst affected countries with over 101,500 confirmed cases and more than 5,696 confirmed deaths at the time of writing (17/9 2020) .1 COVID-19 is caused by the corona virus SARSCoV-2 and presents with a wide spectrum of clinical symptoms. Wu et al reported that 81% of people with COVID-19 in China presented with mild symptoms; 14% presented with symptoms of severe respiratory dysfunction; and 5% developed a critical illness with respiratory failure, septic shock, and multiple organ dysfunction or failure.2 The medium and long-term problems experienced by survivors of COVID-19 after discharge from hospital are currently unknown, but there is some emerging evidence. An Italian study followed-up 143 individuals 7 weeks post-discharge and found 53% reporting fatigue, 43% breathlessness and 27% joint pain.3 Post-discharge symptoms may also be predicted from the previous coronavirus outbreaks of Severe Acute Respiratory Syndrome (SARS) in 2002 and Middle East Respiratory Syndrome (MERS) in 2012. A meta-analysis of 28 follow-up studies found that one quarter of hospitalised survivors of SARS and MERS had reduced lung function and exercise capacity at six months post-discharge.4 At one year, post-traumatic stress disorder (PTSD), depression and anxiety, and reduced quality of life were observed Specific data concerning the rehabilitation needs of this group is therefore urgently required.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed as covid 19 with chest ct and/or nasopharyngeal swab for covid 19
2. age 18 years old and above
3. post covid syndrome after 6 weeks

Exclusion Criteria:

* 1-below age of 18 2 -not confirmed cases 3. symptoms less than 6 weeks

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: will be carried out in Assuit university hospital among health team workers(doctors, nurses, employes), in Emergency room(ER) , clinics , ICU and wards for patients who had covid 19
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Identify post covid symptoms | after 4 weeks of diagnosis
  by interview questionnaire

SECONDARY OUTCOMES:
prevalance of post covid syndrome among survivours | after 4 weeks of diagnosis
  by interview questionnaire

REFERENCES:
- See also: Related Info — https://www.care.gov.eg/EgyptCare/Index.aspx